CLINICAL TRIAL: NCT04457115
Title: Comparison of Efficacy of Ultrasound-guided Erector Spinae Plane Block Versus Thoracic Paravertebral Block for Intra and Postoperative Pain Control in Modified Radical Mastectomy: a Randomized Controlled Trial.
Brief Title: Erector Spinae Plane Block Versus Thoracic Paravertebral Block for Pain Control in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AUSL Romagna Rimini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ELETTRA; 2613 (Registry Identifier: Reg. sperimentazioni)
Record Dates: First submitted 2020-06-22; First posted 2020-07-07 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Breast Surgery; Thoracic Paravertebral Block; Post-operative Pain Control; Erector Spinae Plane Block; Opioid Use
Keywords: breast surgery; Thoracic paravertebral block; Erector spinae plane block; Mastectomy; post-operative pain control

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPV Block (Experimental): Thoracic paravertebral block performed at thoracic level T2-T3 and T4-T5 with administration of Ropivacaine 0.7% 8 ml for each level.
  Interventions: Procedure: Thoracic paravertebral block
- ESP Block (Experimental): Erector spinae plane block performed at thoracic level T2 and T5 with administration of Ropivacaine 0.5% 12 ml for each level.
  Interventions: Procedure: Erector spinae plane Block

INTERVENTIONS:
Procedure: Thoracic paravertebral block — Thoracic paravertebral block performed at T2-T3 and T4-T5 levels with administration of Ropivacaine 0.7% 8 ml for each level
  Arms: TPV Block
Procedure: Erector spinae plane Block — Erector spinae plane block performed at T2 and T5 levels with administration of Ropivacaine 0.5% 12 ml for each level
  Arms: ESP Block

SUMMARY:
The aim of the study is to compare the effectiveness of the Erector spinae plane (ESP) block versus thoracic paravertebral (TPV) block in the post-operative pain control after radical mastectomy.

DETAILED DESCRIPTION:
Primary outcome of our study is to compare the effectiveness of two regional anesthesia techniques, ESP block and TPV block, in the post-operative pain-control after radical mastectomy.

We will also evaluate both intra and post-operative opioid consumption, the incidence of PONV, the length of hospital stay, patient satisfaction with the anesthesiology technique and the incidence of chronic pain 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 85
* American Society of Anesthesiologists classification I - III
* Signature of consent to participate in the study

Exclusion Criteria:

* Coagulopathies and / or use of antiplatelet / anticoagulant drugs
* Infections and/or lesions at the puncture site,
* BMI ≥40
* allergies and / or contraindications to the administration of the drugs used in the study,
* use of chronic opioid therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Post-operative pain assessment | 12 hours
  post-operative pain assessment using Numeric rating scale (from 0,no pain, to 10 ,worst pain)

SECONDARY OUTCOMES:
Length of hospital stay | 3 days
  The number of days of hospitalization after surgery will be assessed
Evaluate the incidence and severity of persistent pain 6 months after surgery | six months
  Evaluate the incidence and severity of persistent pain 6 months after surgery using Numeric rating scale (from 0, no pain, to 10, worst pain)
Opioid use | 36 hours
  Intra and post-operative opioid use
Incidence of PONV | 36 hours
  Incidence of post operative nausea and vomiting (PONV) in the first 36 hours
Assessment of patient satisfaction with the anesthesiological technique | 36 hours
  Patients is requested to fill out a pre-printed sheet on their judgment of the anesthesiological procedure, in which they can express a value from 0 to 5, where 0 indicates "entirely dissatisfied" and 5 indi- cates "very satisfied"

CONTACTS AND LOCATIONS:
Overall Officials: Domenico P Santonastaso, MD, Principal Investigator — AUSL Romagna, M. Bufalini Hospital, Cesena
Locations (1):
- Domenico Pietro Santonastaso, Cesena, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santonastaso DP, de Chiara A, Righetti R, Marandola D, Sica A, Bagaphou CT, Rosato C, Tognu A, Curcio A, Lucchi L, Russo E, Agnoletti V. Efficacy of bi-level erector spinae plane block versus bi-level thoracic paravertebral block for postoperative analgesia in modified radical mastectomy: a prospective randomized comparative study. BMC Anesthesiol. 2023 Jun 16;23(1):209. doi: 10.1186/s12871-023-02157-2. PMID 37328817